CLINICAL TRIAL: NCT01229943
Title: Randomized Phase II Study of Everolimus Alone Versus Everolimus Plus Bevacizumab in Patients With Locally Advanced or Metastatic Pancreatic Neuroendocrine Tumors
Brief Title: Everolimus and Octreotide Acetate With or Without Bevacizumab in Treating Patients With Locally Advanced or Metastatic Pancreatic Neuroendocrine Tumors That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02609; NCI-2011-02609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000687459; CALGB-80701; CALGB-80701 (Other: Alliance for Clinical Trials in Oncology); CALGB-80701 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Advanced Pancreatic Neuroendocrine Tumor; Locally Advanced Pancreatic Neuroendocrine Tumor; Pancreatic Gastrinoma; Pancreatic Neuroendocrine Tumor G1; Pancreatic Neuroendocrine Tumor G2; Pancreatic Vipoma
MeSH Terms: conditions — Vipoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Everolimus; Octreotide; Acetates; Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (octreotide acetate and everolimus) (Experimental): Patients receive 28-day cycles until progression or unacceptable toxicity consisting of: everolimus 10 mg PO QD on days 1-28 and octreotide acetate 20 mg IM on day 1.
  Interventions: Drug: Everolimus; Drug: Octreotide Acetate
- Arm II (octreotide acetate, everolimus, and bevacizumab) (Experimental): Patients receive 28-day cycles until progression or unacceptable toxicity consisting of: everolimus 10 mg PO QD on days 1-28, octreotide acetate 20 mg IM on day 1 and bevacizumab 10 mg/kg IV on days 1 and 15.
  Interventions: Biological: Bevacizumab; Drug: Everolimus; Drug: Octreotide Acetate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
  Arms: Arm II (octreotide acetate, everolimus, and bevacizumab)
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Drug: Octreotide Acetate — Given IM
  Other Names: D-Phenylalanyl-L-cysteinyl-L-phenylalanyl-D-tryptophyl-L-lysyl-L-threonyl-N-[(1R,2R)-2-hydroxy-1-(hyroxymethyl)propyl]-L-cysteinamide, Cyclic (2->7)-disulfide, Acetate (Salt); Longastatin; Longastatina; Samilstin; Sandostatin; Sandostatin Lar Depot; Sandostatina; Sandostatine; SMS 201-995; SMS 201-995 AC

SUMMARY:
This randomized phase II trial studies how well everolimus and octreotide acetate with or without bevacizumab works in treating patients with pancreatic neuroendocrine tumors that cannot be removed by surgery and have spread nearby or to other places in the body. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Octreotide acetate may interfere with and slow the growth of tumor cells. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab and everolimus also may stop the growth of pancreatic neuroendocrine tumors by blocking blood flow to the tumor. It is not yet known whether giving everolimus and octreotide acetate together is more effective with or without bevacizumab in treating pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To assess the progression-free survival rate of patients with locally advanced or metastatic pancreatic neuroendocrine tumors treated with everolimus alone or everolimus plus bevacizumab.

SECONDARY OBJECTIVES:

I. To compare progression-free survival (PFS) among treatment arms shown to be efficacious.

II. To estimate the overall tumor response rate in patients with metastatic pancreatic neuroendocrine tumors treated with one of two novel regimens.

III. To estimate the overall biochemical response rate (as measured by plasma chromogranin A levels) in patients with metastatic pancreatic neuroendocrine tumors treated with these regimens.

IV. To assess the toxicity of each regimen in patients with metastatic pancreatic neuroendocrine tumors.

V. To assess the overall survival of patients with pancreatic neuroendocrine tumors treated with these regimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive everolimus orally (PO) once daily (QD) on days 1-28 and octreotide acetate intramuscularly (IM) on day 1.

ARM II: Patients receive everolimus and octreotide acetate as in Arm I. Patients also receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic documentation of well-differentiated or moderately differentiated neuroendocrine tumor from either a primary or metastatic site

  * If different histologic classification schemes are used, equivalent histologic classifications (for example "grade 1", "low-grade", or "intermediate-grade") are allowed
  * Patients with poorly differentiated neuroendocrine carcinoma or small cell carcinoma are excluded
  * Documentation from a metastatic disease site is sufficient if there is clinical evidence of a pancreatic primary site
* Locally unresectable or metastatic disease
* Patients must have either histologic documentation of a pancreatic primary site, or clinical evidence of a pancreatic neuroendocrine primary tumor as determined by the treating physician

  * Patients with neuroendocrine tumors (e.g., gastrinoma, VIPoma) in whom a pancreatic or peripancreatic primary site is strongly suspected are also eligible
* Patients must have evidence of disease (measurable or non-measurable) with evidence of progression within the past 12 months
* Measurable disease:

Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan

* Non-measurable disease:

All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions; lesions that are considered non-measurable include the following:

* Bone lesions
* Leptomeningeal disease
* Ascites
* Pleural/pericardial effusion
* Inflammatory breast disease
* Lymphangitis cutis/pulmonis
* Abdominal masses that are not confirmed and followed by imaging techniques
* Cystic lesions

  * No prior treatment with bevacizumab, everolimus, or other mammalian target of rapamycin (mTOR) inhibitors
  * Other prior treatments, including but not limited to prior cytotoxic chemotherapy, alpha interferon, tyrosine kinase inhibitors, external beam radiation therapy, and radiopeptide therapy are allowed
* There is no limit on the number of prior treatment regimens
* Any prior treatment (with the exception of octreotide) must be completed at least 4 weeks prior to initiation of treatment

  * Prior treatment with embolization or ablative therapies is allowed if measurable disease remains outside of the treated area
* There is no limit on the prior number of procedures

  * Treatment with somatostatin analogs is a requirement of the study
* Patients receiving octreotide at the time of study entry may continue at the same dose level for the duration of the study
* Patients not receiving octreotide will initiate treatment according to study guidelines
* Prior progression on somatostatin analogs or a negative octreotide scan does not exclude patient participation in this study

  * Patients should have completed any major surgery >= 4 weeks from start of treatment
* Patients must have completed any minor surgery >= 2 weeks prior to start of treatment
* Patients must have fully recovered from the procedure
* Insertion of a vascular access device is not considered major or minor surgery

  * Patients should not receive immunization with attenuated live vaccines within one week prior to registration or during protocol therapy
  * No concurrent condition resulting in immune compromise, including chronic treatment with corticosteroids or other immuno suppressive agents
  * No active or severe liver disease (e.g., acute or chronic hepatitis, cirrhosis); no positive anti-hepatitis B virus (HBV); HBV seropositive patients (hepatitis B surface antigen [HBsAg] positive) are eligible if they are closely monitored for evidence of active HBV infection by HBV deoxyribonucleic acid (DNA) testing, and they agree to receive suppressive therapy with lamivudine or other HBV-suppressive therapy until at least 4 weeks after the last dose of everolimus; patients who are hepatitis C antibody positive are eligible provided that hepatitis C viral load (hepatitis C ribonucleic acid [RNA]) is undetectable
  * No clinical evidence of brain metastases or carcinomatous meningitis
  * No history of gastrointestinal (GI) perforation within 12 months prior to registration
  * No history of clinically significant bleeding episodes
  * Patients on therapeutic anticoagulation are eligible for the study provided that they are on a stable dose of anticoagulants
  * No uncontrolled diabetes mellitus
  * Patients with a history of severely impaired lung function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or oxygen (O2) saturation that is 88% or less at rest on room air are excluded
  * Patients with fasting serum cholesterol >= 300 mg/dL OR >= 7.75 mmol/L AND fasting triglycerides >= 2.5 X upper limit of normal (ULN) should initiate lipid-lowering medications with the goal of achieving levels below these thresholds
  * No history of intolerance or allergies to octreotide
  * Patients with a history of hypertension must be adequately controlled (baseline blood pressure [BP] < 150/90 mm Hg) on antihypertensives
  * No current congestive heart failure (New York Heart Association class II, III, or IV)
  * No symptomatic arterial peripheral vascular disease
  * No history of aortic aneurysm, aortic dissection, angina, myocardial infarction, stroke, or other arterial thrombotic events within 6 months of registration
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-1
  * Women must not be pregnant or lactating; both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study
  * Granulocytes >= 1,500/uL
  * Platelets >= 100,000/uL
  * Creatinine =< 1.5 x upper limit of normal
  * Bilirubin =< 1.5 x upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (=< 5 x upper limit of normal if liver metastases present)
  * Urine protein =< 1+ OR urine creatinine ratio =< 1 (by urinalysis)
* If urine protein creatinine (UPC) ratio is > 1 on urinalysis, then 24-hour urine collection for protein must be obtained and level must be < 1,000 mg for patient enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10-15 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H Kulke, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (394):
- United States (388):
  - Providence Hospital, Mobile, Alabama
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Garnet Health Medical Center, Middletown, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (6):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Vitalite Health Network - Dr Leon Richard Oncology Centre, Moncton, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2010 to October 2012, 150 participants were recruited and randomized to study treatment.
Groups:
- Arm I (Octreotide Acetate and Everolimus): Patients receive 28-day cycles until progression or unacceptable toxicity consisting of: everolimus 10 mg PO QD on days 1-28 and octreotide acetate 20 mg IM on day 1.> > Everolimus: Given PO>
  > Octreotide Acetate: Given IM
- Arm II (Octreotide Acetate, Everolimus, and Bevacizumab): Patients receive 28-day cycles until progression or unacceptable toxicity consisting of: everolimus 10 mg PO QD on days 1-28, octreotide acetate 20 mg IM on day 1 and bevacizumab 10 mg/kg IV on days 1 and 15.>
  > Bevacizumab: Given IV>
  > Everolimus: Given PO>
  > Octreotide Acetate: Given IM
Period: Overall Study
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab)
Started | 75 | 75
Completed | 57 | 58
Not Completed | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Median (Full Range); unit: years] | 59 [23 to 80] | 58 [21 to 86] | 58.5 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 40 | 44 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 69 | 70 | 139
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 8 | 12
  White | 64 | 61 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 6 | 11
  United States | 70 | 69 | 139

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) was defined as the time from study entry until disease progression or death, whichever occurs first. The median PFS was estimated using the Kaplan-Meier method. Progression was assessed per RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions (and an absolute increase of at least 0.5 cm) or the appearance of new lesions.
Time Frame: From study entry to the date of documented progression or death from any cause, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab)
Number analyzed (Participants) | 75 | 75
months | 14.0 [9.1 to 16.9] | 16.7 [12.6 to 19.7]
Statistical Analysis 1: Comparison: Arm I (Octreotide Acetate and Everolimus) vs Arm II (Octreotide Acetate, Everolimus, and Bevacizumab); Based on the log rank test, with 130 patients enrolled over 22 months and followed an additional 24 months, the difference in median PFS between 9 months and 14 months can be detected with approximately 90% power (1-sided, α=0.15); Test type: Superiority or Other; p = 0.12, Log Rank — Tests were stratified by: prior treatment with cytotoxic chemotherapy (no vs yes), prior use of octreotide (no vs yes), and prior therapy with sunitinib (no vs yes); Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.55 to 1.17]

2. Secondary Outcome: Overall Response Rate
Description: The proportion of patients who respond (completely or partially) to each combination regimen will be estimated. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab)
Number analyzed (Participants) | 75 | 75
percentage of participants | 12 | 31

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from study entry to death from any cause. The median OS was estimated using the Kaplan-Meier method.
Time Frame: From registration to time of death, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab)
Number analyzed (Participants) | 75 | 75
months | 35.0 [29.9 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 36.7 [31.8 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

ADVERSE EVENTS:
Description: 147 participants were evaluable for adverse events.
Arm/Group | Arm I (Octreotide Acetate and Everolimus) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 20/74 | 31/73
Other Adverse Events (participants affected / at risk) | 73/74 | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Octreotide Acetate and Everolimus) (N=74) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab) (N=73)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 16 (25)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 4 (5)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 5 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (5)
Bloating (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 14 (18)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 8 (8) | 13 (16)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (12)
Chills (General disorders) | 0 (0) | 2 (4)
Edema limbs (General disorders) | 2 (2) | 11 (15)
Edema trunk (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 15 (18) | 21 (31)
Fever (General disorders) | 2 (2) | 5 (7)
Malaise (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 5 (5)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 2 (2)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (8) | 7 (9)
Alkaline phosphatase increased (Investigations) | 2 (3) | 9 (13)
Aspartate aminotransferase increased (Investigations) | 8 (9) | 12 (20)
Blood bilirubin increased (Investigations) | 1 (2) | 5 (8)
CPK increased (Investigations) | 1 (2) | 0 (0)
Cholesterol high (Investigations) | 4 (4) | 6 (8)
Creatinine increased (Investigations) | 3 (3) | 9 (13)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 4 (5)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (4) | 2 (4)
Neutrophil count decreased (Investigations) | 4 (5) | 2 (2)
Platelet count decreased (Investigations) | 4 (7) | 9 (16)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 3 (4)
Weight loss (Investigations) | 0 (0) | 12 (18)
White blood cell decreased (Investigations) | 0 (0) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 11 (13)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (12) | 21 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 11 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 8 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 7 (8)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 11 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (5)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (4)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 5 (6)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 3 (4)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2) | 13 (17)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 1 (3)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 6 (7) | 18 (26)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Lymphedema (Vascular disorders) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Octreotide Acetate and Everolimus) (N=74) | Arm II (Octreotide Acetate, Everolimus, and Bevacizumab) (N=73)
Anemia (Blood and lymphatic system disorders) | 29 (226) | 40 (332)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (2) | 4 (6)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (7) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (4)
Chest pain - cardiac (Cardiac disorders) | 2 (7) | 1 (3)
Heart failure (Cardiac disorders) | 0 (0) | 2 (12)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 4 (9)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (8)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (21) | 2 (24)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (5)
Tinnitus (Ear and labyrinth disorders) | 2 (37) | 3 (9)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (22)
Blurred vision (Eye disorders) | 4 (36) | 6 (13)
Cataract (Eye disorders) | 0 (0) | 1 (4)
Conjunctivitis (Eye disorders) | 2 (5) | 3 (5)
Dry eye (Eye disorders) | 2 (37) | 4 (30)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 3 (35) | 3 (9)
Eye pain (Eye disorders) | 0 (0) | 1 (2)
Floaters (Eye disorders) | 1 (19) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (4)
Watering eyes (Eye disorders) | 1 (13) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (12) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 26 (115) | 25 (62)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (5)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (2) | 3 (25)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 4 (13) | 10 (27)
Constipation (Gastrointestinal disorders) | 15 (54) | 17 (67)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 48 (244) | 50 (324)
Dry mouth (Gastrointestinal disorders) | 6 (67) | 5 (9)
Dyspepsia (Gastrointestinal disorders) | 9 (65) | 7 (37)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (8) | 2 (3)
Flatulence (Gastrointestinal disorders) | 5 (57) | 11 (37)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 5 (31)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (12) | 4 (14)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3) | 1 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 9 (49)
Ileal fistula (Gastrointestinal disorders) | 0 (0) | 1 (4)
Lip pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 48 (280) | 43 (173)
Nausea (Gastrointestinal disorders) | 36 (158) | 38 (154)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (10) | 3 (11)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (11)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 4 (7)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Toothache (Gastrointestinal disorders) | 2 (3) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 14 (32) | 22 (61)
Chills (General disorders) | 6 (30) | 13 (71)
Dysmenorrhea (General disorders) | 0 (0) | 1 (2)
Edema face (General disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 17 (83) | 25 (175)
Edema trunk (General disorders) | 1 (1) | 1 (3)
Facial pain (General disorders) | 1 (2) | 1 (2)
Fatigue (General disorders) | 60 (521) | 63 (521)
Fever (General disorders) | 9 (14) | 7 (12)
Flu like symptoms (General disorders) | 4 (15) | 5 (11)
Gait disturbance (General disorders) | 2 (6) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 3 (3) | 3 (3)
Localized edema (General disorders) | 2 (2) | 2 (5)
Malaise (General disorders) | 0 (0) | 3 (24)
Neck edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 5 (7)
Pain (General disorders) | 12 (85) | 16 (59)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (5)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (16)
Immune system disorders - Other (Immune system disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 2 (2) | 5 (11)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (22)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (6) | 4 (10)
Skin infection (Infections and infestations) | 5 (8) | 4 (7)
Tooth infection (Infections and infestations) | 3 (3) | 4 (4)
Upper respiratory infection (Infections and infestations) | 7 (14) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (17)
Vulval infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (7)
Bruising (Injury, poisoning and procedural complications) | 2 (7) | 3 (5)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 3 (25)
Intraoperative skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (10)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 28 (158) | 28 (172)
Alkaline phosphatase increased (Investigations) | 22 (126) | 32 (275)
Aspartate aminotransferase increased (Investigations) | 38 (182) | 40 (317)
Blood bilirubin increased (Investigations) | 3 (10) | 9 (33)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 5 (11)
CPK increased (Investigations) | 1 (2) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 29 (178) | 35 (216)
Creatinine increased (Investigations) | 9 (35) | 18 (103)
Hemoglobin increased (Investigations) | 1 (3) | 1 (3)
INR increased (Investigations) | 1 (1) | 3 (17)
Investigations - Other (Investigations) | 2 (9) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (89) | 8 (33)
Lymphocyte count increased (Investigations) | 4 (12) | 1 (2)
Neutrophil count decreased (Investigations) | 26 (74) | 17 (43)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 29 (202) | 34 (198)
Weight gain (Investigations) | 0 (0) | 5 (17)
Weight loss (Investigations) | 17 (73) | 27 (132)
White blood cell decreased (Investigations) | 17 (99) | 14 (76)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 21 (104) | 27 (104)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (25) | 2 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 54 (485) | 56 (479)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (11) | 8 (16)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (6) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 5 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 36 (161) | 37 (249)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (24) | 8 (28)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (44) | 23 (116)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (46) | 25 (89)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (22) | 6 (9)
Hypokalemia (Metabolism and nutrition disorders) | 9 (30) | 16 (53)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (81) | 14 (77)
Hyponatremia (Metabolism and nutrition disorders) | 10 (42) | 18 (76)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (38) | 21 (58)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 4 (10) | 2 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (59) | 11 (111)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (11) | 2 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (78) | 8 (39)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (31) | 10 (58)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (52) | 5 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (88) | 12 (45)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (49) | 11 (33)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 2 (23) | 1 (1)
Dizziness (Nervous system disorders) | 11 (52) | 13 (24)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (9)
Dysgeusia (Nervous system disorders) | 9 (39) | 13 (75)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 23 (120) | 32 (150)
Memory impairment (Nervous system disorders) | 1 (24) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 3 (51) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (5)
Paresthesia (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (35) | 15 (42)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (10)
Agitation (Psychiatric disorders) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (47) | 7 (66)
Confusion (Psychiatric disorders) | 0 (0) | 4 (4)
Delusions (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 7 (88) | 8 (74)
Insomnia (Psychiatric disorders) | 17 (148) | 18 (146)
Libido decreased (Psychiatric disorders) | 1 (11) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (5)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (2) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 8 (45)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 4 (5) | 5 (16)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 3 (41)
Proteinuria (Renal and urinary disorders) | 12 (42) | 46 (393)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 4 (7)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (11) | 4 (44)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (23)
Urinary tract pain (Renal and urinary disorders) | 2 (3) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (22)
Genital edema (Reproductive system and breast disorders) | 1 (2) | 1 (5)
Irregular menstruation (Reproductive system and breast disorders) | 2 (2) | 3 (21)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (22)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (9)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (60) | 18 (47)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (30) | 12 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (37) | 46 (242)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (28)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (18) | 8 (36)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (22)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (60)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 4 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (9) | 4 (39)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (22)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 10 (11)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (25) | 4 (20)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (16) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (60) | 16 (128)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (22) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 3 (35) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (7)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (15) | 2 (4)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (76) | 11 (70)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (32) | 11 (87)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24 (66) | 38 (151)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9 (67) | 11 (131)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (8) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (3) | 1 (8)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 3 (3) | 5 (6)
Hypertension (Vascular disorders) | 38 (226) | 59 (542)
Hypotension (Vascular disorders) | 1 (1) | 4 (5)
Lymphedema (Vascular disorders) | 1 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (9) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less